CLINICAL TRIAL: NCT01392365
Title: Development of a Prediction Model for Differential Diagnosis Between Intestinal Tuberculosis and Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Byong Duk Ye, Associate Professor, Asan Medical Center
Other Study IDs: 2011-0380
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Crohn's Disease; Intestinal Tuberculosis
Keywords: Crohn's disease; Intestinal tuberculosis; Diagnosis, Differential
MeSH Terms: conditions — Crohn Disease; Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Crohn' disease: The group of patients whose final diagnosis is Crohn's disease
- Intestinal tuberculosis: The group of patients whose final diagnosis is intestinal tuberculosis

SUMMARY:
The aim of this study is to develop a scoring system and a prediction model for differential diagnosis between intestinal tuberculosis and Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease and intestinal tuberculosis mimic each other in clinical, endoscopic, and histological features. In addition, the yield of microbiological/histological test (AFB stain, caseating granuloma) is not high in clinical setting. Therefore, distinguishing CD from ITB especially in highly endemic areas for TB is challenging. The aim of this study is to develop and to validate a scoring system and a prediction model for differential diagnosis between intestinal tuberculosis and Crohn's disease

ELIGIBILITY:
Final diagnostic criteria:

* Crohn' disease (at least two of the following is met)

  1. Clinical history of abdominal pain, weight loss, malaise, diarrhea, and/or rectal bleeding
  2. Endoscopic findings of mucosal cobblestoning, linear ulceration, skip areas, or perianal disease
  3. Radiologic findings of stricture, fistula, mucosal cobblestoning, or ulceration
  4. Macroscopic appearance of bowel-wall induration, mesenteric lymphadenopathy, and "creeping fat" at laparotomy
  5. Pathologic findings of transmural inflammation and/or epithelioid granulomas
* Intestinal tuberculosis(at least one of the following is met)

  1. Histologic evidence of caseating granulomas
  2. Histologic demonstration of acid-fast bacilli
  3. Growth of M. tuberculosis on tissue culture
  4. Clinical, colonoscopic, radiologic, and/or operative evidence of Intestinal tuberculosis with proved tuberculosis elsewhere
  5. Response to antituberculous therapy without subsequent recurrence in patients with clinical, colonoscopic, radiologic, and/or operative evidence of Intestinal tuberculosis

Exclusion Criteria:

* Refusal to participate in the study
* Age: 15 years or younger
* Comorbidity with acute infectious disease
* Pregnancy
* Previous history of medication including anti-TB drugs, immunosuppressive drugs, and chemotherapeutic agents\
* Use of antibiotics within the previous three months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected to have intestinal tuberculosis or Crohn's disease based on clinical history, symptoms, and/or colonoscopic findings are invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2011-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Final diagnosis (Intestinal tuberculosis or Crohn's disease) | 6 months (In a subset of patients, for diagnosis of intestinal tuberculosis, final colonoscopic evaluation after completion of 6-months anti-tuberculous medication is needed)
  Patients with suspected diagnosis of intestinal tuberculosis or Crohn's disease will be invited to participate in this study. Study variables including past medical history, clinical symptoms and signs, laboratory variables, radiologic findings (Chest X-ray and small bowel follow-through, colonoscopic features) will be gathered at study enrollment. Final diagnosis of intestinal tuberculosis or Crohn's disease will be made according to the diagnostic criteria previously described (Lee YJ, et al. Endoscopy 2006;38:592-597). A prediction model using various variables for intestinal tuberculosis or Crohn's disease will be constructed in the development group and will be validated in the validation group.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almadi MA, Ghosh S, Aljebreen AM. Differentiating intestinal tuberculosis from Crohn's disease: a diagnostic challenge. Am J Gastroenterol. 2009 Apr;104(4):1003-12. doi: 10.1038/ajg.2008.162. Epub 2009 Feb 24. PMID 19240705
- [Result] Makharia GK, Srivastava S, Das P, Goswami P, Singh U, Tripathi M, Deo V, Aggarwal A, Tiwari RP, Sreenivas V, Gupta SD. Clinical, endoscopic, and histological differentiations between Crohn's disease and intestinal tuberculosis. Am J Gastroenterol. 2010 Mar;105(3):642-51. doi: 10.1038/ajg.2009.585. Epub 2010 Jan 19. PMID 20087333
- [Result] Lee YJ, Yang SK, Byeon JS, Myung SJ, Chang HS, Hong SS, Kim KJ, Lee GH, Jung HY, Hong WS, Kim JH, Min YI, Chang SJ, Yu CS. Analysis of colonoscopic findings in the differential diagnosis between intestinal tuberculosis and Crohn's disease. Endoscopy. 2006 Jun;38(6):592-7. doi: 10.1055/s-2006-924996. Epub 2006 Apr 27. PMID 16673312
- [Derived] Bae JH, Park SH, Ye BD, Kim SO, Cho YK, Youn EJ, Lee HS, Hwang SW, Yang DH, Kim KJ, Byeon JS, Myung SJ, Yang SK. Development and Validation of a Novel Prediction Model for Differential Diagnosis Between Crohn's Disease and Intestinal Tuberculosis. Inflamm Bowel Dis. 2017 Sep;23(9):1614-1623. doi: 10.1097/MIB.0000000000001162. PMID 28682807